CLINICAL TRIAL: NCT01551290
Title: A Phase 3, Multicenter, Randomized, Double-Blind, Placebo-Controlled Study Evaluating the Efficacy and Safety of Infliximab in Chinese Subjects With Active Ulcerative Colitis
Brief Title: A Study to Evaluate the Effectiveness and Safety of Infliximab in Chinese Patients With Active Ulcerative Colitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Xian-Janssen Pharmaceutical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR018769; REMICADEUCO3001 (Other: Xian-Janssen Pharmaceutical Ltd., China)
Record Dates: First submitted 2012-03-07; First posted 2012-03-12 (Estimated); Last update posted 2015-10-30 (Estimated); Status verified 2015-10

CONDITIONS: Ulcerative Colitis
Keywords: Ulcerative colitis; UC; Remicade; Infliximab; Chinese patients; Mayo score; Mucosal healing; Rectal bleeding; Inflammatory bowel disease; IBD
MeSH Terms: conditions — Colitis, Ulcerative; Gastrointestinal Hemorrhage; Inflammatory Bowel Diseases | interventions — Infliximab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group I: Placebo (Placebo Comparator): Participants in Group I receive placebo
  Interventions: Drug: Placebo
- Group II: Infliximab (Experimental): Participants in Group II receive 5 mg/kg infliximab
  Interventions: Drug: Infliximab

INTERVENTIONS:
Drug: Infliximab — Form = solution for injection, route = intravenous (IV), Unit = mg/kg, number = 5, administered on = Weeks 0, 2, 6, 14, and 22 and for extension phase: participants treated with infliximab through Week 22 will receive infliximab at Weeks 30, 38, 46 and 54, and will receive placebo at Week 32 and 34.
  Arms: Group II: Infliximab
Drug: Placebo — Form = solution for injection, route = IV, administered on = Weeks 0, 2, 6, 14, and 22 and for extension phase: participants treated with placebo through Week 22 will receive infliximab at Weeks 32, 34, 38, 46 and 54 and will receive placebo at Week 30.
  Arms: Group I: Placebo

SUMMARY:
The purpose of this study is to evaluate the effectiveness and safety of infliximab in Chinese patients with active ulcerative colitis (swelling and ulceration of large intestine and rectum).

DETAILED DESCRIPTION:
This is a multicenter (study conducted at multiple sites), randomized (the study medication is assigned by chance), placebo controlled (placebo is an inactive substance that is compared with a medication to test whether the medication has a real effect in a clinical study), double blind (neither investigator nor patient knows the treatment that the patient receives), 2-arm (2 groups), parallel group (a clinical study comparing the response in two or more groups of participants receiving different treatments) study with infliximab in patients with active ulcerative colitis. The study consists of screening period (4 weeks prior to baseline [patient's medical status before any treatment or research is done] at Week 0), treatment period (Week 0 to Week 22) and follow up period (Week 26). Participants completing treatment till Week 22 and benefit from continued treatment (in the opinion of the investigator) may enter a study extension period from Week 30 until Week 58. Hundred participants will be randomized to 2 groups: Group 1 (50 participants receiving placebo) and Group 2 (50 participants receiving infliximab). Effectiveness and safety (physical examination, and a review of AEs, vital signs, laboratory analyses, and concomitant medications) will be evaluated at Week 8 and Week 26 and at Week 58 (for participants who enter extension phase). The maximum duration for participants in the main study is 26 weeks. The maximum duration for participants including study extension is 58 weeks. One of the specialized procedures used to calculate efficacy will be Mayo score which is calculated using the subscore (recorded in Mayo Diary Card by each participant) of the following 4 variables (1) stool frequency (scores ranging from 0 [normal number stools for this patient] to 3 [5 or more stools more than normal]), (2) rectal bleeding (scores ranging from 0 [no blood seen] to 3 [blood alone passed]), (3) endoscopic findings (scores ranging from 0 [normal or inactive disease] to 3 [severe disease ie, spontaneous bleeding and ulceration]), and (4) the physician's global assessment (scores ranging from 0 [normal] to 3 [severe disease]).

ELIGIBILITY:
Inclusion Criteria:

* Has active ulcerative colitis of at least 3 months duration at screening with score of ≥2 on the endoscopy subscore of the Mayo score and baseline Mayo score of 6 to 12
* Concomitant medications: either have concurrent treatment with at least 1 of the therapies (eg, oral corticosteroids and 6-Mercaptopurine [6-MP]).
* Has to be eligible according to the tuberculosis (TB) eligibility assessment

Exclusion Criteria:

* Has severe extensive colitis or ulcerative colitis limited to only the rectum or to less than 20 cm of the colon
* Requires or required within 2 months prior to screening any surgery for active gastrointestinal bleeding, peritonitis (inflammation of abdominal lining), intestinal obstruction, or intra-abdominal or pancreatic abscess (a localized collection of pus in pancreas) requiring surgical drainage -Has severe fixed symptomatic stenosis (narrowing of the opening or hollow of any passage) of large or small intestine
* Has colonic obstruction or history within the 6 months prior to baseline
* Has colonic mucosal dysplasia (colonic mucosal cell maturation abnormality) or its history
* Has a history of extensive colonic resection (extensive partial removal of colon), lymphoproliferative disease (disease in which lymphocytes are produced in excessive quantities), demyelinating disease (disease of the nervous system)
* Has adenomatous colonic polyps (benign projecting mass of large intestine), stoma (opening either natural or surgically created connecting a portion of the body cavity to the outside environment), known infection of Human immunodeficiency virus (HIV), hepatitis B and C
* Has had treatment with cyclosporine, tacrolimus, sirolimus, or mycophenolate mofetil within 8 weeks prior to screening

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2012-04; Primary Completion 2014-03 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Number of participants with a clinical response at Week 8 | Week 8
  At Week 8, clinical response is defined as a decrease from baseline (closest measurement taken prior to or at the time of the initiation of the baseline [Week 0] infusion) in the Mayo score by ≥30% and ≥3 points, with a decrease in the rectal bleeding subscore of ≥1 or a rectal bleeding subscore of 0 or 1, at Week 8.

SECONDARY OUTCOMES:
Number of participants in clinical remission at Week 8 | Week 8
  A clinical remission at Week 8 is defined as a Mayo score ≤2 points, with no individual subscore >1. Participants in remission by this definition will have rectal bleeding subscore of either 0 or 1.
Number of participants with mucosal healing at Week 8 | Week 8
  Mucosal healing is determined from the endoscopy subscore of the Mayo score. Mucosal healing will be defined by endoscopy subscore of 0 or 1.
Number of participants with a clinical response at Week 26 | Week 26
  At Week 26, clinical response is defined as decrease from baseline in the Mayo score by ≥30% and ≥3 points, with a decrease in the rectal bleeding subscore of ≥1 or a rectal bleeding subscore of 0 or 1, at Week 26.
Number of participants in clinical remission at Week 26 | Week 26
  A clinical remission at Week 26 is defined as a Mayo score ≤2 points, with no individual subscore >1. Participants in remission by this definition will have rectal bleeding subscore of either 0 or 1.

CONTACTS AND LOCATIONS:
Overall Officials: Xian-Janssen Pharmaceutical Ltd. Clinical Trial, Study Director — Xian-Janssen Pharmaceutical Ltd.
Locations (7):
- China (7):
  - Beijing
  - Chengdu
  - Guangzhou
  - Hefei
  - Shanghai
  - Wuhan
  - Xi'an

REFERENCES:
- See also: A Phase 3, Multicenter, Randomized, Double-Blind, Placebo-Controlled Study Evaluating the Efficacy and Safety of Infliximab in Chinese Subjects With Active Ulcerative Colitis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_7051&studyid=3324&filename=REMICADEUCO3001-Synopsis.pdf